CLINICAL TRIAL: NCT00408655
Title: Phase I Study of CCI-779 (NSC 683864) in Combination With Carboplatin and Paclitaxel in Patients With Advanced Solid Tumours
Brief Title: Temsirolimus, Carboplatin, and Paclitaxel in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00691; NCI-2009-00691 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000652060; IND.179 (Other: National Cancer Institute of Canada Clinical Trials Group); NCIC-179 (Other: CTEP)
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Ovarian Sarcoma; Ovarian Stromal Cancer; Recurrent Endometrial Carcinoma; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Stage III Endometrial Carcinoma; Stage III Ovarian Epithelial Cancer; Stage III Ovarian Germ Cell Tumor; Stage IV Endometrial Carcinoma; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Endometrial Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; Taxes; Carboplatin; temsirolimus; Sirolimus

ARMS (1):
- Arm I (Experimental): PART A: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30-60 minutes on day 1 and temsirolimus IV over 30 minutes on days 8 and 15. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  PART B: Patients receive paclitaxel and carboplatin as in part A. They also receive temsirolimus IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: temsirolimus

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
This phase I trial is studying the side effects and best dose of temsirolimus, carboplatin, and paclitaxel in treating patients with advanced solid tumors. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving temsirolimus together with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and recommended phase II dose of temsirolimus, carboplatin, and paclitaxel in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. Determine the frequency and severity of toxic effects of this regimen in these patients.

II. Document any evidence of objective antitumor activity of this regimen in patients with measurable disease.

III. Determine the pharmacokinetic profile of carboplatin and paclitaxel alone, temsirolimus alone, and carboplatin, paclitaxel, and temsirolimus in combination in these patients.

OUTLINE: This is a multicenter, open-label, dose-escalation study. Patients receive treatment in either part A or part B.

PART A: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 30-60 minutes on day 1 and temsirolimus IV over 30 minutes on days 8 and 15. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

PART B: Patients receive paclitaxel and carboplatin as in part A. They also receive temsirolimus IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients in parts A and B receive escalating doses of temsirolimus, carboplatin, and paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The recommended phase II dose (RPTD) is the dose that is one dose level below the MTD. Once the RPTD is determined in part A, patients are enrolled in part B. An expanded cohort of up to 10 patients with endometrial or ovarian cancer are treated at the RPTD determined in part B (final RPTD).

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Criteria:

* Histologically confirmed solid tumors
* Measurable or nonmeasurable disease: No serum tumor marker elevation as the only evidence of disease; Patients with ovarian or endometrial cancer must have measurable disease, defined as >= 1 lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Advanced disease; Refractory to standard therapy OR no standard therapy is available
* Carboplatin and paclitaxel considered reasonable therapeutic option
* No known brain metastases
* ECOG performance status 0-1
* Life expectancy >= 12 weeks
* Absolute granulocyte count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT =< 3 times ULN (5 times ULN if documented liver metastases)
* Fasting serum cholesterol =< 9.0 mmol/L
* Fasting triglycerides =< 4.56 mmol/L
* Creatinine normal OR creatinine clearance >= 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Accessible for treatment and follow up
* No serious cardiovascular illness, including any of the following:

myocardial infarction within the past 6 months, congestive heart failure (even if medically controlled), unstable angina, active cardiomyopathy, cardiac arrhythmia, uncontrolled hypertension

* No preexisting sensory or motor neuropathy >= grade 2 due to previous chemotherapy; Local or regional neurological findings related to previous injury or disease allowed
* No hearing loss >= grade 2 from any cause
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to temsirolimus
* No serious illness or medical condition that would preclude study treatment including, but not limited to, any of the following: History of significant neurologic or psychiatric disorder that would impair the ability to obtain consent or limit study compliance, Active uncontrolled infection or nonhealing wounds, OR;
* At least 4 weeks since prior radiotherapy (except low-dose, palliative radiotherapy) and recovered
* At least 4 weeks since prior chemotherapy and recovered
* No more than 2 prior chemotherapy regimens
* Prior therapy with carboplatin and/or paclitaxel allowed provided the patient has no persistent related toxicity >= grade 1 AND retreatment with the combination is clinically indicated (e.g., second-line therapy for ovarian cancer with > 6-month treatment-free interval)
* At least 21 days since prior major surgery and recovered
* No prior mTOR inhibitor
* No concurrent prophylactic hematopoietic colony-stimulating factors
* No other concurrent anticancer therapy or investigational agents
* Active peptic ulcer disease, Any other medical condition that might be aggravated by treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-02; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose of temsirolimus, carboplatin, and paclitaxel | Up to 3 years
Safety | Up to 3 years
Tolerability | Up to 3 years
Dose-limiting toxicities | Up to 3 years

SECONDARY OUTCOMES:
Efficacy | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada